CLINICAL TRIAL: NCT05319652
Title: Co-development and Assessment of the Feasibility and Potential Effects of an Online Self-management Program for Chronic Non-cancer Pain
Brief Title: Feasibility Study of an Online Self-management Program for Chronic Non-cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Anne-Marie-Pinard, Anesthesiologist, CHU de Quebec-Universite Laval
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-6312
Record Dates: First submitted 2022-03-21; First posted 2022-04-08 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain self-management program (Experimental): Participants log in to the online program and develop practical strategies to manage CNCP.
  Interventions: Behavioral: Pain self-management program

INTERVENTIONS:
Behavioral: Pain self-management program — Each week for eight weeks, participants are invited to complete self-directed lessons on particular themes. The program covers goal setting, stress management through relaxation, breathing and mindfulness, pacing, physical activity, thoughts and emotions, sleep, nutrition, flare-up management, and planning. Through pain education, positive testimonials from individuals with CNCP applying the suggested strategies, reflective activities, goal setting and monitoring, and the gradual development of a personal plan, the program supports self-efficacy building to manage CNCP.

SUMMARY:
Based on a mixed-methods design, the objective of this trial is to assess the feasibility and acceptability of the "Agir pour moi" program, an 8-week online self-management program for chronic non-cancer pain (CNCP). The investigators will also explore its potential effects on self-efficacy, pain interference, pain severity, anxiety, depression, catastrophizing, and global impression of change in adults with CNCP awaiting services from a chronic pain multidisciplinary treatment center.

DETAILED DESCRIPTION:
The mixed-methods sequential explanatory design combines a quantitative questionnaire-based study with a subsequent in depth qualitative approach.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* live with CNCP for more than 3 months;
* read and understand French easily;
* have access to a computer and high-speed Internet;
* be available to take part in the project for 6 to 8 months;
* not having started a new treatment for pain within the last month;
* agree to notify the team before starting a new treatment;
* be able to give informed consent.

Exclusion Criteria:

* be supported by a multidisciplinary treatment center or be likely to be in the short term;
* having participated in a CNCP self-management program within the last year;
* be awaiting scheduled surgical treatment within six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of the recruitment | Baseline
  * Number of potentially eligible adults referred by the multidisciplinary treatment center over the recruitment period
  * Number of referred adults who respond to the invitation
  * Number of referred adults who consent to participate in the study
  * Number of interested adults excluded based on inclusion/exclusion criteria
Feasibility of data collection | Baseline
  * Rate of response to the questionnaires
  * Rate of completed questionnaires (no missing data)
Feasibility of data collection | Post-intervention (8 weeks)
  * Rate of response to the questionnaires
  * Rate of completed questionnaires (no missing data)
Feasibility of data collection | 3 months post-intervention
  * Rate of response to the questionnaires
  * Rate of completed questionnaires (no missing data)
Acceptability | Post-intervention (8 Weeks)
  The Acceptability E-scale includes 6 items regarding how easy and enjoyable the program was to use, how understandable were the lessons, how helpful was completing the program, whether the participant liked the program, whether the amount of time to complete the program was acceptable, and overall satisfaction with the program. Scores can range from 6 to 30. Higher scores reprensent a high level of acceptability.
Acceptability | 4 months post-intervention
  Qualitative data from semi-structured interviews
Adherence to the program | Post-intervention (8 weeks)
  Completion rate of the program (completion is following ≥ 75% of the lessons)

SECONDARY OUTCOMES:
Change in self-efficacy: French version of the Pain Self-Efficacy Questionnaire (PSEQ) | Baseline; Post-intervention (8 weeks); 3 months post-intervention
  The PSEQ is a ten item questionnaire which assesses an individual's confidence in their ability to perform a variety of activities or tasks despite pain. Scores can range from 0 to 60. Higher scores represent lower confidence to function with pain.
Change in pain severity and pain interference: French version of the Brief Pain Inventory (BPI) | Baseline; Post-intervention (8 weeks); 3 months post-intervention
  The BPI includes a pain severity subscale and a pain interference subscale. The pain interference subscale measures the extent to which pain interferes with functions such as general activity, walking ability, normal work, mood, relationships with people, enjoyment of life and sleep. For each scale, the total score is the average of all items. Scores can range from 0 to 10 for each subscale. Higher scores indicate greater severity and more interference.
Change in anxiety and depression: French version of the Hospital Anxiety and Depression Scale (HADS) | Baseline; Post-intervention (8 weeks); 3 months post-intervention
  The HADS is a 14-item scale. Seven items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Change in pain catastrophizing: French version of the Pain Catastrophizing Scale (PCS) | Baseline; Post-intervention (8 weeks); 3 months post-intervention
  The PCS is a 13-item questionnaire designed to assess catastrophic thinking in relation to pain. It yields a total score and three subscale scores assessing rumination, magnification and helplessness. Scores can range from 0 to 52. Higher scores represent higher pain catastrophizing.
Patient Global Impression of Change Scale (PGIC) | Post-intervention (8 weeks); 3 months post-intervention
  The PGIC measures a patient's rating of overall improvement or lack thereof due to the intervention. It is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Pinard, MD, M(Ed.), Principal Investigator — CHU de Quebec-Universite Laval
Locations (1):
- CHU de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marier-Deschenes P, Pinard AM, Jalbert L, LeBlanc A. Assessing the Feasibility and Preliminary Effects of a Web-Based Self-Management Program for Chronic Noncancer Pain: Mixed Methods Study. JMIR Hum Factors. 2024 May 3;11:e50747. doi: 10.2196/50747. PMID 38701440